CLINICAL TRIAL: NCT06559254
Title: Randomized Controlled Trial of Transcranial Direct Current Stimulation (tDCS) as Augmentation Therapy to Cognitive Training (CT) in Individuals With Major Neurocognitive Disorder (MND) of Mild Severity
Brief Title: TDCS as Augmentation Therapy to Cognitive Training in Mild Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Ying, Resident, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 24-305
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Major Neurocognitive Disorder
Keywords: mild dementia; major neurocognitive disorder; tdcs; transcranial direct current stimulation; cognitive training
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tdcs with cognitive training (Active Comparator): active transcranial direct current stimulation with cognitive training by N-back using computerized programme
  Interventions: Device: transcranial direct current stimulation
- Sham tdcs with cognitive training (Sham Comparator): Sham transcranial direct current stimulation with cognitive training by N-back using computerized programme
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation by applying weak current through electrode. It can archive excitation by anode stimulation or inhibition by stimulating cathode. By inducing modification of membrane polarisation, it can modulate cerebral excitability. Literature suggested anode tDCS over the dorsolateral prefrontal cortex (DLPFC) improved cognitive function, in terms of responding faster and more accurate in cognitive tasks. tDCS was well tolerated and accepted by participants.

SUMMARY:
Due to increase in life expectancy, major neurocognitive disorder (MND) becoming increasingly important as reflected in the increasing number in dementia population, as well as in burden to health care system and to caregiver.

Among current treatment, cognitive training has shown to have significant outcome in cognitive impaired patient. But the effect is reported to be small and might not be long-lasting. In consideration of the neuronal excitability effect in tDCS, it may consolidate the effect of cognitive training if used simultaneously. The study will investigate on efficacy of tDCS as combined intervention to cognitive training.

The study aims to investigate the efficacy of 2-week (5 sessions per week) tDCS to augment cognitive training in subjects with MND with clinically mild severity. Patients with diagnosis of MND or dementia from HKWC will be recruited with inclusion and exclusion criteria listed. The eligible participants will be randomized to receive either active intervention (active tDCS) or sham (sham tDCS) as control with cognitive training simultaneously.

Each session lasts for 20 minutes. The subjects will be allocated to either interventional or control group using block randomization. Block of 4 will be used to allocate subjects at 1:1 ratio between two groups. Both the participants and investigators responsible for assessment and data analysis will be blinded to the group allocation. Primary and secondary outcome will be assessed at baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention. Baseline assessment assesses on demographic data (e.g. age, gender, years of education), clinical data with full psychiatric assessment and access to previous medical record, neuropsychiatric data (HK-MoCA and CNPI). Primary outcomes includes N-back (cognitive training) performance, forward and backward digit span. Secondary outcomes includes measurement on dementia rating and trail making test. In data analysis, any group differences in demographics and clinical profiles between the intervention and sham group at baseline will be assess. ANOVA will be performed to examine the effect of time and intervention on primary outcome and other cognitive assessment across time points. Potential confounders will be adjusted.

Baseline assessments and outcome measures is either psychiatric assessment, clinician rating scales or cognitive assessment performed with investigator.

DETAILED DESCRIPTION:
Due to increase in life expectancy, major neurocognitive disorder (MND) becoming increasingly important as reflected in the increasing number in dementia population, as well as in burden to health care system and to caregiver.

Among current treatment, cognitive training has shown to have significant outcome in cognitive impaired patient. But the effect is reported to be small and might not be long-lasting. In consideration of the neuronal excitability effect in tDCS, it may consolidate the effect of cognitive training if used simultaneously. The study will investigate on efficacy of tDCS as combined intervention to cognitive training.

The study aims to investigate the efficacy of 2-week (5 sessions per week) tDCS to augment cognitive training in subjects with major neurocognitive disorder with clinically mild severity. Patients with diagnosis of MND or dementia from HKWC will be recruited with inclusion and exclusion criteria listed. The eligible participants will be randomized to receive either active intervention (active tDCS) or sham (sham tDCS) as control with cognitive training simultaneously.

Each session lasts for 20 minutes. The subjects will be allocated to either interventional group or control group using block randomization. Block of 4 will be used to allocate subjects at 1:1 ratio between two groups. Both the participants and investigators responsible for assessment and data analysis will be blinded to the group allocation. Primary outcome and secondary outcome will be assessed at baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention. Baseline assessment assesses on demographic data (e.g. age, gender, years of education), clinical data with full psychiatric assessment and access to previous medical record, neuropsychiatric data (HK-MoCA and CNPI). Primary outcomes includes N-back (cognitive training) performance, forward and backward digit span. Secondary outcomes includes measurement on dementia rating and trail making test. In data analysis, any group differences in demographics and clinical profiles between the intervention and sham group at baseline will be assess. ANOVA will be performed to examine the effect of time and intervention on primary outcome and other cognitive assessment across time points. Potential confounders will be adjusted.

Baseline assessments and outcome measures is either psychiatric assessment, clinician rating scales or cognitive assessment performed with investigator. No questionnaires will be given to participants.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or above
* Right-handedness Chinese as defined by Edinburgh handedness inventory
* Cantonese speaking
* Fulfil the criteria of Major neurocognitive disorder, as defined by the 5 th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM- 5)
* Clinical Dementia Rating Global score = 1

Exclusion Criteria:

* Active diagnosis of mood disorder or psychosis
* Alcohol or substance dependence
* Initiation or change in dose of cognitive enhancer within 6 months prior to the onset of the study 14
* Poor physical condition and mobility
* Having regular cognitive training (as defined by at least three 1-hour weekly structured and standardized cognitive training in recent 3 months) 15
* Receiving tDCS within 2 months prior to the onset of study 16
* Significant communication or visual impairment
* Having metal implant in area above upper back, or having metal crown or metal brace, or pacemaker

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
N-back task performance in terms of reaction time and % of correct | Baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention
  N-back task performance in terms of reaction time and % of correct. The data will be measured in the computerized programme.
Forward and Backward digit span | Baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention
  Digit span is widely used to test verbal working memory. It can be assessed in forward (forward digit span) and reverse order (backward digit span). It is also a component in Wechsler Adult Intelligence Scale.

SECONDARY OUTCOMES:
Clinical dementia rating - sum of boxes | Baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention
  Clinical dementia rating (CDR) is a 5-point scale to assess six domains of cognitive and functional performance. The Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) has increased utility in detecting difference between stages of dementia severity.
Chinese version of the neuropsychiatric inventory (CNPI) | Baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention
  CNPI is developed by Cummings et al. It assesses 12 aspects in neuropsychiatric disturbances, e.g. agitation, anxiety, irritability. The modified version of NPI also evaluate carer distress.
Trail making test | Baseline, week 2 (after course of intervention) and 4 weeks after the course of intervention
  Trail Making Test (TMT) is widely used test to assess attention, psychomotor speed and mental flexibility. Trail making test - black and white (TMT-B&W) used numbers in circle with black and white background instead of use of the English alphabet in Trail Making Test part B (TMT B). It is more user friendly in individuals would might not be able to read English letters.

CONTACTS AND LOCATIONS:
Overall Officials: Pak Wing Cheng, MBBS, HKU, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Need to further liase with hospital authority over data share for research purpose.

REFERENCES:
- [Background] Kim HJ, Baek MJ, Kim S. Alternative type of the trail making test in nonnative English-speakers: the trail making test-black & white. PLoS One. 2014 Feb 13;9(2):e89078. doi: 10.1371/journal.pone.0089078. eCollection 2014. PMID 24551221
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Cruz Gonzalez P, Fong KNK, Chung RCK, Ting KH, Law LLF, Brown T. Can Transcranial Direct-Current Stimulation Alone or Combined With Cognitive Training Be Used as a Clinical Intervention to Improve Cognitive Functioning in Persons With Mild Cognitive Impairment and Dementia? A Systematic Review and Meta-Analysis. Front Hum Neurosci. 2018 Oct 16;12:416. doi: 10.3389/fnhum.2018.00416. eCollection 2018. PMID 30386223
- [Background] Lampit A, Hallock H, Suo C, Naismith SL, Valenzuela M. Cognitive training-induced short-term functional and long-term structural plastic change is related to gains in global cognition in healthy older adults: a pilot study. Front Aging Neurosci. 2015 Mar 9;7:14. doi: 10.3389/fnagi.2015.00014. eCollection 2015. PMID 25805989
- [Background] Jones RW. Have cholinergic therapies reached their clinical boundary in Alzheimer's disease? Int J Geriatr Psychiatry. 2003 Sep;18(Suppl 1):S7-S13. doi: 10.1002/gps.936. PMID 12973745
- [Background] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Background] Mintun MA, Lo AC, Duggan Evans C, Wessels AM, Ardayfio PA, Andersen SW, Shcherbinin S, Sparks J, Sims JR, Brys M, Apostolova LG, Salloway SP, Skovronsky DM. Donanemab in Early Alzheimer's Disease. N Engl J Med. 2021 May 6;384(18):1691-1704. doi: 10.1056/NEJMoa2100708. Epub 2021 Mar 13. PMID 33720637
- [Background] Tricco AC, Ashoor HM, Soobiah C, Rios P, Veroniki AA, Hamid JS, Ivory JD, Khan PA, Yazdi F, Ghassemi M, Blondal E, Ho JM, Ng CH, Hemmelgarn B, Majumdar SR, Perrier L, Straus SE. Comparative Effectiveness and Safety of Cognitive Enhancers for Treating Alzheimer's Disease: Systematic Review and Network Metaanalysis. J Am Geriatr Soc. 2018 Jan;66(1):170-178. doi: 10.1111/jgs.15069. Epub 2017 Sep 29. PMID 29131306